CLINICAL TRIAL: NCT00102921
Title: Pilot, Double-Blind, Placebo-Controlled, Parallel Group Study of the Safety Clinical Activity of CCX282-B in Patients With Moderate to Severe Crohn's Disease
Brief Title: Safety and Activity Study of an Oral Medication to Treat Moderate to Severe Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL003_282
Record Dates: First submitted 2005-02-04; First posted 2005-02-07 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; oral medication
MeSH Terms: conditions — Crohn Disease | interventions — CCX282-B

INTERVENTIONS:
Drug: CCX282-B

SUMMARY:
The purpose of this research study is to investigate the effects of an investigational medication, called CCX282-B, on safety and on the some of the symptoms of Crohn's Disease in patients who are experiencing an active flare-up of moderate to severe Crohn's Disease.

DETAILED DESCRIPTION:
CCX282-B is being developed as a treatment for inflammatory bowel diseases such as Crohn's Disease. CCX282-B is a highly potent, orally active, chemokine receptor antagonist whose single target is the G-protein coupled receptor CCR9. The CCR9 receptor is expressed by most T-cells in the thymus as well as in the intestine, and by a small population of T-cells in the peripheral blood. In humans, the CCR9 receptor is implicated in Crohn's Disease and ulcerative colitis.

Crohn's Disease is an autoimmune disease involving the entire length of the gastrointestinal tract, but with most manifestations in the terminal small intestine and colon. This condition is characterized by mucosal ulcerations that penetrate deeply into the bowel wall. Sometimes the ulcerative lesions completely penetrate the bowel wall, leading to fistula formation and infectious complications requiring surgical intervention. Patients experience considerable lifestyle disruption and disability from this disease, including diarrhea, abdominal pain, malnutrition, anemia, and repetitive surgeries to remove disease-affected gastrointestinal segments.

ChemoCentryx Protocol CL003_282 is a double-blind, placebo-controlled, parallel group, two stratum, Phase 2A pilot study of the safety, tolerability, immunologic and clinical activity, and population pharmacokinetics of a single dose level of CCX282-B administered daily for four consecutive weeks to patients with active, moderate to severe Crohn's Disease. The primary immunologic and clinical activity objective of this study is to provide pilot information regarding the immunologic and clinical activity of daily oral doses of CCX282-B in the treatment of moderate to severe Crohn's Disease, based on changes in the Crohn's Disease Activity Index (CDAI). Secondary immunologic and clinical activity objectives include evaluation of the effect of CCX282-B on the Inflammatory Bowel Disease Questionnaire (IBDQ) instrument, C-reactive protein (CRP), the endoscopic appearance and biopsy of the colon and terminal ileum, and markers of leukocyte subsets and activation status. The primary safety objective of this study is to evaluate the safety and tolerability of oral doses of CCX282-B in patients with moderate to severe Crohn's Disease. In addition, blood samples will be collected for evaluation of the population pharmacokinetics of CCX282-B.

Study acquired by Amgen and all disclosures were done by previous sponsor ChemoCentryx.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe Crohn's Disease in small intestine; disease must be active at the time of study entry
* Use of adequate and approved methods of birth control throughout the study period
* Willing and able to sign an informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Infection with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV; the virus that causes AIDS)
* Abuse of alcohol or of illegal drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2004-08; Study Completion 2005-12

PRIMARY OUTCOMES:
Crohn's Disease Activity Index score
Safety (Adverse Events, tolerability)

SECONDARY OUTCOMES:
Inflammatory Bowel Disease Questionnaire
C-reactive protein
Endoscopic appearance and biopsy of colon and terminal ileum
Markers of leukocyte subsets and activation status

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (14):
- United States (14):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Rocky Mountain Clincal Research, Golden, Colorado
  - Arapahoe Gastroenterology, Littleton, Colorado
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Long Island Clinical Research Associates, LLP, Great Neck, New York
  - Wake Forest Research, Raleigh, North Carolina
  - University Hospitals of Cleveland, Div of Gastroenterology, Cleveland, Ohio
  - Digestive Disease Clinic, Jackson, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Center for Colon Rectal Disease, Salt Lake City, Utah
  - University of Virginia Health System, Digestive Health Center of Excellence, Charlottesville, Virginia